CLINICAL TRIAL: NCT03623451
Title: Serum Metabolomics Study of Traditional Chinese Medicine Formula （Shen Qi Tiao Ti Formula） Intervention to Polycystic Ovary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yan Li, Clinical professor, Heilongjiang University of Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shen Qi Tiao Ti_PCOS
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chinese Medicine Formula (Experimental): All 100 patients were treated with Chinese Medicine Formula(CMF) for three menstrual cycles.
  Interventions: Drug: Chinese Medicine Formula

INTERVENTIONS:
Drug: Chinese Medicine Formula — Chinese Medicine Formula, composed of American ginseng 10g, Poria cocos 15g, bighead atractylodes rhizome 20g, Astragalus mongholicus 30g, Crataegus pinnatifida Bunge 20g, Salvia miltiorrhiza Bge. 20g, Pericarpium Citri Reticulatae 10g will be decocted and packaged into vacuum packs by the pharmaceutical department of First Affiliated Hospital, Heilongjiang University of Chinese Medicine (140 mL/pack). Subjects will take 2 packages per day for three months.

SUMMARY:
Polycystic ovary syndrome (PCOS) is a most common, heterogeneous, complex endocrinopathy disease.Traditional Chinese medicine (TCM) has been used in the treatment of PCOS for many years. However, the mechanism underlying TCM remains obscure and challenging.In the present study, a metabolomics approach based on ultra-high-performance liquid chromatography (UPLC) coupled with linear ion trap Orbi-trap mass spectrometer (LTQ Orbi-trap MS) is used to investigate serum metabolic changes of TCM intervention to PCOS.

ELIGIBILITY:
Inclusion Criteria:

* PCOS diagnostic criteria: According to the diagnostic criteria revised by the European Society of Human Reproduction and Embryology and the American Society for Reproductive Medicine at the Rotterdam in 2003, PCOS patients can be diagnosed if two of the three criteria are present after excluding congenial adrenal hyperplasia, Cushing's syndrome, androgen secreting tumors, or other related disorders. The three criteria are (1) oligo- and/or anovulation; (2) clinical and/or biochemical signs of hyperandrogenism (clinical manifestations of hyperandrogenism include presence of acne, hirsutism, and androgenic alopecia); (3) polycystic ovaries by ultrasound examination: presence of 12 or more follicles in each ovary measuring 2-9 mm on diameter and/or ovarian volume>10 ml.
* Age between 14 and 40 years.
* 2 years after menarche

Exclusion Criteria:

* Administration of other medications known to affect reproductive function or metabolism within the past three months, including oral contraceptives, Gonadotropin-releasing hormone (GnRH) agonists and antagonists, anti androgens, gonadotropins, anti-obesity drugs, Chinese herbal medicines, anti diabetic drugs such as metformin and thiazolidinediones, somatostatin, diazoxide, and calcium channel blockers.
* Patients with other endocrine disorders including 21-hydroxylase deficiency, hyperprolactinemia, uncorrected thyroid disease, suspected Cushing's syndrome.
* Patients with known severe organ dysfunction or mental illness.

Ages: 14 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
The fatty acid amides (FAAs) metabolite changes | 3 months
  The metabolic changes before and after treatment

SECONDARY OUTCOMES:
The sulfated steroids metabolite changes | 3 months
  The metabolic changes before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided